CLINICAL TRIAL: NCT02200328
Title: Efficacy of Metronidazole Prophylaxis Against Clostridium Difficile-Associated Diarrhea in High Risk Adult Patients: A Randomized Clinical Trial
Brief Title: Efficacy of Metronidazole Prophylaxis Against Clostridium Difficile-Associated Diarrhea in High Risk Adult Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patients noncompliant with instructions and follow ups could not be completed.
Sponsor: Alison Schneider (Other)
Responsible Party: Sponsor-Investigator, Alison Schneider, M.D, Cleveland Clinic Florida
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLA14-061
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Clostridium Difficile Diarrhea
Keywords: Clostridium difficile infection; Diarrhea; Flagyl; Metronidazole
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Metronidazole; Starch

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Experimental): Metronidazole tablets 500mg orally or IV , 3 times a day for a maximum of 14 days
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Placebo(Corn starch pill) orally 3 times a day for a maximum of 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — Metronidazole tablets 500mg orally or IV , 3 times a day for a maximum of 14 days
  Other Names: Flagyl
  Arms: Metronidazole
Drug: Placebo — Placebo(Corn starch pill) orally 3 times a day for a maximum of 14 days
  Other Names: corn starch pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to test if metronidazole prophylaxis is effective in decreasing the incidence of hospital induced Clostridium Difficile diarrhea among patients at high risk for this infection.

DETAILED DESCRIPTION:
Clostridium Difficile infection or C. Diff (CDI) is an infection that causes severe diarrhea. Risk factors for this infection include hospitalization, the use of antibiotics, along with medications that decrease the acid in the stomach. This infection leads to a disease which is difficult to treat and can cause serious complications including death in rare cases. This infection also increases medical costs by prolonging hospital stays.

Metronidazole (known by the brand name Flagyl) is an antibiotic that has been available for decades and has been used to treat this disease. Flagyl is approved by the Food and Drug Administration for the treatment of C. diff infection. Recent research by the investigators group has shown that hospitalized patients who took Flagyl had a decreased chance of getting C. Diff infection. However, high quality studies are needed to better evaluate whether the investigators can prevent C. Diff infection in high risk patients with the use of Flagyl.

The purpose of this study is to assess if metronidazole prophylaxis is effective in decreasing the incidence of hospital induced Clostridium Difficile diarrhea among inpatients at high risk for this infection.

High risk patient population are as defined below: taking a broad spectrum antibiotics (piperacillin/tazobactam-Zosyn; Ciprofloxacin).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients >55
* Proton Pump inhibitor / Histamine-2 Blocker
* On broad spectrum antibiotics (Zosyn and/or Ciprofloxacin). These two antibiotics are selected based on current hospital formulary/use
* Anticipated hospital stay >48 hours
* Mental capacity (able to give informed written consent).

Exclusion Criteria:

* Admission for CDI
* Existing diarrhea at admission
* Passed prophylactic window (>48 hours on broad spectrum antibiotics)
* Unable to take PO at the time of evaluation for study entry
* No more than 14 days of broad spectrum antibiotics anticipated
* Medications with serious interactions/contraindications to that would be taken together with metronidazole (ex. Warfarin, disulfiram, phenytoin, calcineurin inhibitors)
* Inflammatory Bowel Disease
* Admission for colonic bowel surgery or h/o total/Subtotal colectomy)
* Hospice
* Mortality expected <7days
* Previous CDI in the past 6 months
* Intensive care admission due to the difficulty of monitoring them
* Allergy to Metronidazole or other Antibiotics in protocol
* Patients with neuropathy
* History of heavy ethyl alcohol intake(greater than 3 drinks daily) or intake in past 24 hours,Solid organ transplant.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Schneider, M.D., Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metronidazole | Placebo
Started | 43 | 33
Completed | 0 | 0
Not Completed | 43 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole | Placebo | Total
Number analyzed (Participants) | 43 | 33 | 76
Age, Continuous [Mean (Full Range); unit: years] | 71 [55 to 96] | 71.8 [58 to 98] | 71.4 [55 to 98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 25 | 19 | 44
Region of Enrollment [Number; unit: participants]
  United States | 43 | 33 | 76

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Clostridium Difficile Diarrhea in Both Study Groups at 30 Days Post Broad Spectrum Antibiotic Use.
Time Frame: 30 days
Population: 0 participants were analyzed due to large number of patients not complying to the instructions and loss to follow up.
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Determine Differences in Clostridium Difficile Diarrhea Incidence Between Patients on Piperacillin/Tazobactam vs. Patients on Ciprofloxacin.
Time Frame: 30 days
Population: 0 participants were analyzed due to large number of patients not complying to the instructions and loss to follow up.
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Metronidazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/33
Other Adverse Events (participants affected / at risk) | 0/43 | 0/33

LIMITATIONS AND CAVEATS:
Early termination:

1. Many patients did not comply with the protocol instructions.
2. Lack of resources to conduct the study.
3. Many patients did not respond to follow up calls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes